CLINICAL TRIAL: NCT02063152
Title: 102 Annual Pap Smear Screening Database Maintenance Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201305072RINC
Record Dates: First submitted 2014-02-10; First posted 2014-02-14 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Cancer; Human Papillomavirus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years

GROUPS / COHORTS (1):
- Entire Taiwan women

SUMMARY:
This study aimed to evaluate the subsequent cancer risks, including gynecological cancers and malignancies at other sites, after the detection of screening positives and the diagnosis for primary cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Citizens in Taiwan
* Women who attended screening, or who were diagnosed as cervical cancer
* Women who did not attend screening for at least 6 years

Exclusion Criteria:

* Women died before the follow-up initiation
* Women who had received hysterectomy before the follow-up initiation

Ages: 20 Years to 130 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women attended screening and found abnormal results, and women who were diagnosed as cervical cancer were the main study population. Women who did not attend screening for at least 6 years were also included.
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 1995-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Time to the cancer diagnosis or the recurrence, the death, or the last date of follow-up, whichever came first | up to 25 years

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — Department of Obstetrics and Gynecology, College of Medicine, National Taiwan University
Locations (1):
- Taiwan Cervical Cancer Prevention Monitoring Center, Taipei, Taiwan

REFERENCES:
- [Derived] Tai YJ, Chen YY, Hsu HC, Chiang CJ, You SL, Chen CA, Cheng WF; Taiwan Cervical Cancer Control Task Force. Risks of cervical intraepithelial neoplasia grade 3 or invasive cancers in ASCUS women with different management: a population-based cohort study. J Gynecol Oncol. 2018 Jul;29(4):e55. doi: 10.3802/jgo.2018.29.e55. Epub 2018 Mar 20. PMID 29770625